CLINICAL TRIAL: NCT02782104
Title: An Open-label Long-term Extension Safety Study of Esketamine Nasal Spray in Treatment-resistant Depression
Brief Title: A Long-term Safety Study of Esketamine Nasal Spray in Treatment-resistant Depression
Acronym: SUSTAIN-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108149; 54135419TRD3008 (Other: Janssen Research & Development, LLC); 2015-003578-34 (EudraCT Number)
Record Dates: First submitted 2016-04-29; First posted 2016-05-25 (Estimated); Results first posted 2024-02-20 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Treatment-Resistant
Keywords: Depressive Disorder, Treatment-Resistant; Esketamine; JNJ-54135419
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Esketamine Nasal Spray (Experimental): Open-Label Induction Phase: Participants will self-administer with esketamine nasal spray twice per week for 4 weeks as a flexible dose regimen (56 milligram [mg] or 84 mg for those < 65 years; 28 mg, 56 mg or 84 mg for those >= 65 years). Participants >= 65 years old will start at a dose of 28 mg on Day 1. Optimization/Maintenance Phase: Participants entering from studies ESKETINTRD3001 (NCT02417064), ESKETINTRD3002 (NCT02418585), ESKETINTRD3003 (NCT02493868), ESKETINTRD3004 (NCT02497287), or ESKETINTRD3006 (US sites only) will self-administer esketamine nasal spray (same dose) once weekly. Participants entering from study ESKETINTRD3005 (NCT02422186) will self-administer esketamine nasal spray (28 mg in week 1; 28 or 56 mg in week 2; and 28, 56 or 84 mg in week 3 and 4) once weekly. After Week 4 (starting at Week 5), based on the Investigator's clinical judgment, the dose of esketamine for all participants can be adjusted based upon efficacy and tolerability.
  Interventions: Drug: Esketamine Nasal Spray

INTERVENTIONS:
Drug: Esketamine Nasal Spray — Open-Label Induction Phase: Participants will self-administer with esketamine nasal spray twice per week for 4 weeks as a flexible dose regimen (56 milligram [mg] or 84 mg for those < 65 years; 28 mg, 56 mg or 84 mg for those >= 65 years). Participants >= 65 years old will start at a dose of 28 mg on Day 1. Optimization/Maintenance Phase: Participants entering from studies ESKETINTRD3001 (NCT02417064), ESKETINTRD3002 (NCT02418585) or ESKETINTRD3006 (US sites only) will self-administer esketamine nasal spray (same dose) once weekly. Participants entering from study ESKETINTRD3005 (NCT02422186) will self-administer esketamine nasal spray (28 mg in week 1; 28 or 56 mg in week 2; and 28, 56 or 84 mg in week 3 and 4) once weekly. After Week 4 (starting at Week 5), based on the Investigator's clinical judgment, the dose of esketamine for all participants can be adjusted based upon efficacy and tolerability.
  Other Names: JNJ-54135419

SUMMARY:
The purpose of this study is to assess the safety and tolerability of esketamine nasal spray in participants with treatment-resistant depression (TRD).

DETAILED DESCRIPTION:
This is an open-label (the researchers and participants know the treatment the participant is receiving) long-term extension study. The study will consist of 2 open-label Phases: 4-week Induction phase (if applicable) and Open-Label Optimization/Maintenance phase (variable). Participants will enter the study Induction Phase from ESKETINTRD3001 (NCT02417064), ESKETINTRD3002 (NCT02418585), ESKETINTRD3003 (NCT02493868), ESKETINTRD3005 (NCT02422186) and ESKETINTRD3006 (US sites only). Participants will enter the study Open-Label Optimization/Maintenance phase from ESKETINTRD3001 (NCT02417064), ESKETINTRD3002 (NCT02418585), ESKETINTRD3003 (NCT02493868) (if appropriate at week 16) or ESKETINTRD3006 (US sites only). In the Open-Label Induction Phase, participants will self-administer flexibly-dosed esketamine nasal spray. During first 4 weeks in Optimization/Maintenance Phase responder participants from the induction phase of study 54135419TRD3008, will continue on the same dose of esketamine nasal spray from the induction phase and have a weekly intranasal treatment session frequency. Participants entering the optimization/maintenance phase from study ESKETINTRD3005 will also have a weekly intranasal treatment session frequency. However, as the ESKETINTRD3005 intranasal study medication is blinded at the time of entry into the current study, the dose of esketamine nasal spray will be administered as outlined in protocol. Participants entering the optimization/maintenance phase from study ESKETINTRD3003 (Direct Entry) or ESKETINTRD3004 who were ongoing in the Optimization, Maintenance, or Optimization/Maintenance phase, respectively, will have the option to have their current intranasal dosing frequency adjusted at the time of entry into 54135419TRD3008 study and should remain on the selected frequency from week 1 to week 4. A one-time dose change will be permitted at study entry. After 4 weeks, esketamine nasal spray treatment sessions will be individualized to either once weekly or once every other week at the fixed 2-week interval (based on clinical global impression - severity [CGI-S] performed at that visit), and every 4 weeks for participants dosed at the 4 week interval. Participants safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Based on the prior study the participant is entering 54135419TRD3008 from: a) From ESKETINTRD3001 (NCT02417064) or ESKETINTRD3002 (NCT02418585) study: Participant has completed the induction phase and the 2-weeks follow up phase visit; or Participants completed the induction phase and was a responder and study ESKETINTRD3003 is terminated.; b) From ESKETINTRD3003 (NCT02493868) study: (1) Participant relapsed during the maintenance phase; or (2) Participant was in the induction phase of the ESKETINTRD3003 study when the study was terminated and, after completion of the induction phase, was determined to be a responder; or (3) Participant was in the optimization or maintenance phases at the time the study was terminated; or (4) or (5) Participants was in the induction phase and after completion of induction phase was determined to not meet response criteria (1) Participant completed ESKETINTRD3004 study (optimization/maintenance phase); or (2) Participant was in the induction phase of the ESKETINTRD3004 study when the study was terminated and, after completion of the induction phase, was determined to be a responder; or (3) Participant was in the optimization/maintenance phase at the time the study was terminated; (4) Participant was in the induction phase and did not meet criteria for response may be eligible for to be rolled over into 54135419TRD3008. d) From ESKETINTRD3005 (NCT02422186) study: Participant was in the induction phase of the ESKETINTRD3005 study at the time enrollment into the ESKETINTRD3004 study was closed and, after completion of the induction phase, was determined to be a responder or did not meet the criteria for response. e) From ESKETINTRD3006 study (US Study sites only) (1) Participant completed the induction phase and was a responder.
* Participant must be medically stable on the basis of physical examination, vital signs, pulse oximetry, and 12-lead Electrocardiogram (ECG) performed predose on the day of the first intranasal treatment session. If there are any abnormalities that are not specified in the inclusion and exclusion criteria, their clinical significance must be determined by the investigator and recorded in the participant's source documents and initialed by the investigator
* Participant must be medically stable according to the investigator's judgment and knowledge of the subject's medical stability in the parent study. This determination must be documented.
* A woman of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [b-hCG]) predose on the day of the first intranasal treatment session
* During the study (that is, from the first intranasal treatment session) and for a minimum of 1 spermatogenesis cycle (defined as approximately 90 days) after receiving the last dose of intranasal study medication, a man who is sexually active with a woman of childbearing potential must be practicing a highly effective method of contraception with his female partner c) must agree not to donate sperm.

Exclusion Criteria:

* The evaluation of the benefit versus risk of continued esketamine nasal spray treatment is not favorable for the participant in the opinion of the investigator
* Since the last study visit in the participant's prior study, participant has suicidal ideation with intent to act per the investigator's clinical judgment or based on the Columbia Suicide Severity Rating Scale (C-SSRS) [corresponding to a response of "Yes" on Item 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) in the suicidal ideation module of the C-SSRS] or suicidal behavior per the investigator's clinical judgment or based on the C-SSRS (corresponding to any score higher than 0 in the suicidal behavior module of the C-SSRS)
* Participant has positive test result(s) for drugs of abuse (including barbiturates, methadone, opiates, cocaine, phencyclidine, and amphetamine/methamphetamine) predose on the day of the first intranasal treatment session
* Participant has any anatomical or medical condition that, per the investigator's clinical judgment based on assessment, may impede delivery or absorption of intranasal study drug
* Participant has taken any prohibited therapies that would not permit administration of the first intranasal treatment session

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1148 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (173):
- United States (51):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Garden Grove, California
  - Glendale, California
  - Oakland, California
  - Orange, California
  - San Diego, California
  - San Rafael, California
  - Hartford, Connecticut
  - New Haven, Connecticut
  - Gainesville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Joliet, Illinois
  - Maywood, Illinois
  - Skokie, Illinois
  - Iowa City, Iowa
  - Wichita, Kansas
  - Lake Charles, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Gaithersburg, Maryland
  - Boston, Massachusetts
  - New Bedford, Massachusetts
  - Watertown, Massachusetts
  - Worcester, Massachusetts
  - Rochester Hills, Michigan
  - O'Fallon, Missouri
  - Saint Charles, Missouri
  - Omaha, Nebraska
  - Cedarhurst, New York
  - New York, New York
  - Staten Island, New York
  - Hickory, North Carolina
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Allentown, Pennsylvania
  - Media, Pennsylvania
  - Philadelphia, Pennsylvania
  - Lincoln, Rhode Island
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Wichita Falls, Texas
  - Charlottesville, Virginia
  - Waukesha, Wisconsin
- Argentina (6):
  - Banfield
  - Buenos Aires
  - Córdoba
  - La Plata
  - Mendoza
  - Rosario
- Australia (3):
  - Caulfield
  - Elizabeth Vale
  - Frankston
- Vienna, Austria
- Belgium (6):
  - Aalst
  - Bruges
  - Brussels
  - Heusden-Zolder
  - Liège
  - Yvoir
- Brazil (9):
  - Belo Horizonte
  - Curitiba
  - Fortaleza
  - Passo Fundo
  - Porto Alegre
  - Recife
  - Rio de Janeiro
  - São Bernardo do Campo
  - São Paulo
- Bulgaria (8):
  - Burgas
  - Kardzhali
  - Pazardzhik
  - Pleven
  - Plovdiv
  - Rousse
  - Sofia
  - Varna
- Canada (4):
  - Vancouver, British Columbia
  - Kingston, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
- Czechia (3):
  - Brno
  - Pilsen
  - Prague
- Estonia (2):
  - Tallinn
  - Tartu
- Kuopio, Finland
- France (7):
  - Clermont-Ferrand
  - Douai
  - Nantes
  - Nîmes
  - Paris
  - Poitiers
  - Toulon
- Germany (6):
  - Berlin
  - Bochum
  - Mainz
  - Mittweida
  - Oranienburg
  - Pfaffenhofen
- Hungary (7):
  - Budapest
  - Debrecen
  - Győr
  - Pécs
  - Sopron
  - Szekszárd
  - Vác
- Kaunas, Lithuania
- Kuala Lumpur, Malaysia
- Mexico (6):
  - Guadalajara
  - León
  - Mexico City
  - México
  - Monterrey
  - San Luis Potosí City
- Poland (7):
  - Bełchatów
  - Bialystok
  - Bydgoszcz
  - Gdansk
  - Leszno
  - Lublin
  - Warsaw
- Slovakia (5):
  - Bratislava
  - Liptovský Mikuláš
  - Rimavská Sobota
  - Rožňava
  - Svidník
- South Africa (3):
  - Cape Town
  - Pretoria
  - Welgemoed
- South Korea (2):
  - Gwangju
  - Seoul
- Spain (13):
  - Alcorcón
  - Barcelona
  - Bilbao
  - Madrid
  - Oviedo
  - Palma
  - Pamplona
  - Sabadell
  - Salamanca
  - Sant Boi de Llobregat
  - Torrevieja
  - Vitoria-Gasteiz
  - Zamora
- Sweden (4):
  - Halmstad
  - Lund
  - Skövde
  - Stockholm
- Taiwan (5):
  - Kaohsiung City
  - New Taipei City
  - Taichung
  - Taipei
  - Taoyuan District
- Turkey (Türkiye) (7):
  - Adana
  - Ankara
  - Bursa
  - Istanbul
  - Kucukcekmece/Istanbul
  - Oanakkale
  - Samsun
- United Kingdom (5):
  - Chesterfield
  - Derby
  - London
  - Northampton
  - Oxford

REFERENCES:
- [Derived] Zaki N, Chen LN, Lane R, Doherty T, Drevets WC, Morrison RL, Sanacora G, Wilkinson ST, Young AH, Lacerda ALT, Paik JW, Popova V, Fu DJ. Safety and efficacy with esketamine in treatment-resistant depression: long-term extension study. Int J Neuropsychopharmacol. 2025 Jun 6;28(6):pyaf027. doi: 10.1093/ijnp/pyaf027. PMID 40319349
- [Derived] Castro M, Wilkinson ST, Al Jurdi RK, Petrillo MP, Zaki N, Borentain S, Fu DJ, Turkoz I, Sun L, Brown B, Cabrera P. Efficacy and Safety of Esketamine Nasal Spray in Patients with Treatment-Resistant Depression Who Completed a Second Induction Period: Analysis of the Ongoing SUSTAIN-3 Study. CNS Drugs. 2023 Aug;37(8):715-723. doi: 10.1007/s40263-023-01026-3. Epub 2023 Aug 9. PMID 37558912
- [Derived] Zaki N, Chen LN, Lane R, Doherty T, Drevets WC, Morrison RL, Sanacora G, Wilkinson ST, Popova V, Fu DJ. Long-term safety and maintenance of response with esketamine nasal spray in participants with treatment-resistant depression: interim results of the SUSTAIN-3 study. Neuropsychopharmacology. 2023 Jul;48(8):1225-1233. doi: 10.1038/s41386-023-01577-5. Epub 2023 May 12. PMID 37173512
- [Derived] Starr HL, Abell J, Larish A, Lewis S, DeMuro C, Gogate J, Jamieson C, Daly E, Zaki N, Kramer M. Self-reported review of the value of esketamine in patients with treatment-resistant depression: Understanding the patient experience in the STRIVE Study. Psychiatry Res. 2020 Nov;293:113376. doi: 10.1016/j.psychres.2020.113376. Epub 2020 Aug 8. PMID 32818917

RESULTS

PARTICIPANT FLOW:
Groups:
- Esketamine Nasal Spray: Participants who entered induction phase (IND) from studies NCT02417064, NCT02418585, NCT02493868, NCT02497287, NCT02422186, or ESKETINTRD3006 received esketamine nasal spray twice per week on Day 1 for 4 weeks as a flexible dose regimen (56 milligrams [mg] or 84 mg for participants less than [<] 65 years; 28 mg, 56 mg or 84 mg for participants greater than or equal to [>=] 65 years). Participants who entered the optimization and maintenance phase (OP/MA) from the IND phase of study NCT02782104 continued on the same dose of esketamine from the IND phase, weekly. Participants who entered from studies NCT02417064, NCT02418585, NCT02493868, NCT02497287, or ESKETINTRD3006 were administered esketamine nasal spray, 56 mg or 84 mg, once weekly. Participants who entered from study NCT02422186 received esketamine nasal spray (28 mg in Week 1; 28 or 56 mg in Week 2; and 28, 56 or 84 mg in Weeks 3 and 4) once weekly in OP/MP.
Period: Overall Study
Arm/Group | Esketamine Nasal Spray
Started | 1148
IND Phase (Participants From Study NCT02417064:132; NCT02418585: 51; NCT02493868: 245; NCT02497287: 12; NCT02422186: 3; ESKETINTRD3006: 15) | 458
OP/MA Phase (690 Participants From Study (NCT02417064:0; NCT02418585: 0; NCT02493868: 224; NCT02497287: 455; NCT02422186: 1; ESKETINTRD3006: 10) and 420 Participants from IND Phase) | 1110
Completed | 680
Not Completed | 468
Not completed — Other | 215
Not completed — Induction Day 28 Non Responder | 9
Not completed — Non-Compliance with Study Drug | 2
Not completed — Death | 8
Not completed — Pregnancy | 6
Not completed — Withdrawal by Subject | 63
Not completed — Protocol Violation | 7
Not completed — Lack of Efficacy | 61
Not completed — Lost to Follow-up | 23
Not completed — Adverse Event | 74

BASELINE CHARACTERISTICS:
Arm/Group | Esketamine Nasal Spray
Number analyzed (Participants) | 1148
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 764
  Male | 384
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 200
  Not Hispanic or Latino | 922
  Unknown or Not Reported | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 45
  Black or African American | 45
  Native Hawaiian or Other Pacific Islander | 0
  White | 996
  More than one race | 10
  Unknown or Not Reported | 22
  Other | 29
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 71
  AUSTRALIA | 16
  AUSTRIA | 4
  BELGIUM | 18
  BRAZIL | 100
  BULGARIA | 50
  CANADA | 15
  CZECH REPUBLIC | 90
  ESTONIA | 9
  FINLAND | 1
  FRANCE | 23
  GERMANY | 13
  HUNGARY | 20
  ITALY | 8
  LITHUANIA | 2
  MALAYSIA | 9
  MEXICO | 46
  POLAND | 101
  SLOVAKIA | 9
  SOUTH AFRICA | 48
  SOUTH KOREA | 7
  SPAIN | 41
  SWEDEN | 65
  TAIWAN | 22
  TURKEY | 24
  UNITED KINGDOM | 8
  UNITED STATES | 328

OUTCOME MEASURES:

1. Primary Outcome: Change From Study Baseline in Computerized Cognitive Battery Domain Score: Detection Test (DET) Score
Description: This battery is a series of computerized cognition tests (detection, identification, one card learning, one back and groton maze learning) designed to measure reaction time, visual learning and memory, and executive function/sequencing. The DET is a measure of psychomotor function and uses a well-validated simple reaction time. In this outcome measure, speed of performance of subjects (calculated as mean of the logarithmic base 10 transformed reaction times) for correct responses was reported. Total score ranged from 2 to 3.3 log 10 milliseconds (msec). Lower score indicated better performance. Higher change from baseline indicated better performance.
Time Frame: IND Phase: Baseline up to 4 weeks; OP/MA Phase: Baseline up to 78 months
Population: All enrolled analysis set included all participants who were eligible to enter this study and received at least 1 dose of intranasal study medication. Here, 'N' (number analyzed) signifies number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: log10 msec
Groups:
- Esketamine Nasal Spray (IND Phase): Participants who entered induction phase (IND) from studies NCT02417064, NCT02418585, NCT02493868, NCT02497287, NCT02422186, or ESKETINTRD3006 received esketamine nasal spray twice per week on Day 1 for 4 weeks as a flexible dose regimen (56 milligrams [mg] or 84 mg for participants less than [<] 65 years; 28 mg, 56 mg or 84 mg for participants greater than or equal to [>=] 65 years).
- Esketamine Nasal Spray (OP/MA Phase): Participants who entered the OP/MA phase from the IND phase of study NCT02782104, continued on the same dose of esketamine from the IND phase, weekly. Participants who entered from studies NCT02417064, NCT02418585, NCT02493868, NCT02497287, or NCT02782104 were administered esketamine nasal spray, 56 mg or 84 mg, once weekly. Participants who entered study NCT02422186 received esketamine nasal spray (28 mg in Week 1; 28 or 56 mg in Week 2; and 28, 56 or 84 mg in Weeks 3 and 4) once weekly in optimization and maintenance phase (OP/MP). After Week 4 (starting at Week 5), based on the Investigator's clinical judgment, the dose of esketamine for all participants was adjusted based upon efficacy and tolerability.
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
Number analyzed (Participants) | 420 | 1085
log10 msec | 0.0218 (0.10516) | -0.0065 (0.13526)

2. Primary Outcome: Change From Study Baseline in Computerized Cognitive Battery Domain Score: Identification Test (IDN) Score
Description: This battery is a series of computerized cognition tests (detection, identification, one card learning, one back and groton maze learning) designed to measure reaction time, visual learning and memory, and executive function/sequencing. IDN test is a measure of visual attention (choice reaction time) and scored for speed of response (mean of the log10 transformed reaction times for correct responses). Total score ranged from 2 to 3.3 log 10 msec. Lower score indicated better performance. Higher change from baseline indicated better performance.
Time Frame: IND Phase: Baseline up to 4 weeks; OP/MA Phase: Baseline up to 78 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 msec
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
Number analyzed (Participants) | 422 | 1084
log10 msec | 0.0074 (0.07819) | -0.0185 (0.09893)

3. Primary Outcome: Change From Study Baseline in Computerized Cognitive Battery Domain Score: One Card Learning Test (OCL) Score
Description: This battery is a series of computerized cognition tests (detection, identification, one card learning, one back and groton maze learning) designed to measure reaction time, visual learning and memory, and executive function/sequencing. OCL test is a measure of visual episodic memory and visual recall test scored using arcsine transformation of the percentage of correct responses (CR). The range for OCL is 0 to 100 percent (%) accuracy; presented as an arcsin transformation, the range is 0 to 1.57. Higher score indicated better performance. Higher change from baseline indicated better performance.
Time Frame: IND Phase: Baseline up to 4 weeks; OP/MA Phase: Baseline up to 78 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Arcsine (sqrt of percentage of CR)
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
Number analyzed (Participants) | 429 | 1084
Arcsine (sqrt of percentage of CR) | 0.0170 (0.12356) | 0.0397 (0.15364)

4. Primary Outcome: Change From Study Baseline in Computerized Cognitive Battery Domain Score: One Back Test (ONB) Score
Description: The ONB is a measure of working memory and scored for speed of correct response (mean of the log10-transformed reaction times for correct responses). Total score ranged from 2 to 3.54 log10 msec. Lower score indicated better performance. Higher change from baseline indicated better performance.
Time Frame: IND Phase: Baseline up to 4 weeks; OP/MA Phase: Baseline up to 78 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 msec
Groups:
- Esketamine Nasal Spray (OP/MA Phase): Participants who entered the OP/MA phase from the IND phase of study NCT02782104, continued on the same dose of esketamine from the IND phase, weekly. Participants who entered from studies NCT02417064, NCT02418585, NCT02493868, NCT02497287, or NCT02782104 administered esketamine nasal spray, 56 mg or 84 mg, once weekly. Participants who entered study NCT02422186 were received esketamine nasal spray (28 mg in Week 1; 28 or 56 mg in Week 2; and 28, 56 or 84 mg in Weeks 3 and 4) once weekly in optimization and maintenance phase (OP/MP). After Week 4 (starting at Week 5), based on the Investigator's clinical judgment, the dose of esketamine for all participants was adjusted based upon efficacy and tolerability.
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
Number analyzed (Participants) | 429 | 1084
log10 msec | 0.0086 (0.08096) | 0.0198 (0.10329)

5. Primary Outcome: Change From Study Baseline in Computerized Cognitive Battery Domain Score: Groton Maze Learning Test (GMLT) Score
Description: This battery is a series of computerized cognition tests (detection, identification, one card learning, one back and groton maze learning) designed to measure reaction time, visual learning and memory, and executive function/sequencing. GMLT measures executive function; maze/sequencing test, scored for total number of errors. Total score ranged from 0 to 999 number of errors. Lower score indicated better performance. Higher change from baseline indicated better performance.
Time Frame: IND Phase: Baseline up to 4 weeks; OP/MA Phase: Baseline up to 78 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Errors
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
Number analyzed (Participants) | 415 | 1072
Number of Errors | 1.5 (17.80) | 5.1 (22.52)

6. Primary Outcome: Change From Study Baseline in Hopkins Verbal Learning Test-Revised (HVLT-R) Score
Description: The HVLT-R measures performance in verbal memory, learning, and long-term recall in which a list of words is read up to three times. Approximately 20-25 minutes later, a delayed recall trial and a recognition trial are completed. The delayed recall requires free recall of any words remembered. The recognition trial is composed of 24 words, including the 12 target words and 12 false-positives. When scoring the HVLT, the three learning trials are combined to calculate a total recall score (0-36); the delayed recall trial creates the delayed recall score (0-12); the total number of true-positive errors (0-12); and the range of recognition discrimination index is comprised by subtracting the total number of false positives from the total number of true positives. A higher total recall score indicated higher cognition. The range of the recognition discrimination index is -12 to 12. Higher score indicated better performance and higher change from baseline indicated better performance.
Time Frame: IND Phase: Baseline up to 4 weeks; OP/MA Phase: Baseline up to 78 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
Number analyzed (Participants) | 444 | 1091
score on a scale
  Total Recall | -0.1 (4.05) | 0.8 (5.05)
  Delayed Recall: number analyzed (Participants) | 439 | 1091
  Delayed Recall | 0.3 (3.81) | 0.3 (2.03)
  Total Number of True Positives: number analyzed (Participants) | 443 | 1091
  Total Number of True Positives | 0.1 (2.54) | -0.0 (2.70)
  Recognition Discrimination Index: number analyzed (Participants) | 443 | 1091
  Recognition Discrimination Index | -0.1 (2.88) | -0.1 (3.10)

7. Primary Outcome: Percentage of Participants Based on Columbia-Suicide Severity Rating Scale (C-SSRS) Score
Description: C-SSRS: interview-based instrument to systematically assess suicidal ideation (SI) and behavior, to assess whether participant experienced any of following: completed suicide, suicide attempt (response of "yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior ("yes" on "preparatory acts or behavior", "aborted attempt" or "interrupted attempt"), suicidal ideation ("yes" on "wish to be dead", "non-specific active suicidal thoughts", "active SI with methods without intent to act or some intent to act, without or with specific plan and intent), any self-injurious behavior with no suicidal intent ("yes" on "has participant engaged in non-suicidal self-injurious behavior"). Here, percentage of participants with >=1 positive behavior, participants with >=1 positive ideations; no event were reported.
Time Frame: IND Phase: Baseline up to 4 weeks; OP/MA Phase: Baseline up to 78 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
Number analyzed (Participants) | 456 | 1109
Percentage of participants
  Baseline: No Event | 79.8 | 94.8
  Baseline: Suicidal ideation | 20.2 | 5.2
  Baseline: Suicidal behavior | 0 | 0
  Most Severe Post Baseline: No Event | 77.4 | 70.2
  Most Severe Post Baseline: Suicidal ideation | 22.6 | 27.8
  Most Severe Post Baseline: Suicidal behavior | 0 | 2.0

8. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Any AE occurring at or after the initial administration of study intervention up to end of study was considered as treatment-emergent.
Time Frame: IND Phase: up to 4 weeks; OP/MA Phase: up to 78 months
Population: All enrolled analysis set included all participants who were eligible to enter this study and received at least 1 dose of intranasal study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
Number analyzed (Participants) | 458 | 1110
Participants | 346 | 1052

9. Primary Outcome: Change From Baseline in Heart Rate
Description: Change from baseline (predose) in heart rate were reported.
Time Frame: IND Phase: Baseline up to 4 weeks; OP/MA Phase: Baseline up to 78 months
Population: Full analysis set included participants who received at least 1 dose of intranasal study medication in this study.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
Number analyzed (Participants) | 458 | 1110
beats per minute | 0.4 (9.52) | 0.8 (10.47)

10. Primary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure
Description: Change from baseline in systolic and diastolic blood pressure were reported.
Time Frame: IND Phase: Baseline up to 4 weeks; OP/MA Phase: Baseline up to 78 months
Population: Full analysis set included participants who received at least 1 dose of intranasal study medication in this study.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
Number analyzed (Participants) | 458 | 1110
Millimeters of mercury (mmHg)
  Systolic Blood Pressure | 0.4 (10.72) | 5.8 (12.68)
  Diastolic Blood Pressure | 0.3 (7.47) | 2.7 (8.78)

11. Primary Outcome: Change From Baseline in Respiratory Rate
Description: Change from baseline in respiratory rate were reported.
Time Frame: IND Phase: Baseline up to 4 weeks; OP/MA Phase: Baseline up to 78 months
Population: Full analysis set included participants who received at least 1 dose of intranasal study medication in this study.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
Number analyzed (Participants) | 458 | 1110
breaths per minute | -0.1 (2.51) | -0.4 (2.83)

12. Primary Outcome: Change From Baseline in Blood Oxygen Saturation
Description: Change from baseline in blood oxygen saturation (predose) were reported.
Time Frame: IND Phase: Baseline up to 4 weeks; OP/MA Phase: Baseline up to 78 months
Population: Full analysis set included participants who received at least 1 dose of intranasal study medication in this study.
Measure: Mean (Standard Deviation); unit: percentage of SpO2
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
Number analyzed (Participants) | 458 | 1110
percentage of SpO2 | -0.1 (1.54) | -0.1 (1.63)

13. Secondary Outcome: Change From Baseline in Montgomery Asberg Depression Rating Scale (MADRS) Total Score
Description: MADRS measures depression severity, detects changes due to AD treatment. It consists of 10 items (evaluate apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, suicidal thoughts), scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), summed for a total possible score of 0 to 60. Higher scores indicate more severe conditions. Negative change in score indicates improvement. Missing data was imputed using last observation carried forward (LOCF) method.
Time Frame: IND Phase: Baseline up to 4 weeks; OP/MA Phase: Baseline up to 78 months
Population: Full analysis set included all participants who received at least 1 dose of intranasal study medication in this study. Here, 'N' (number analyzed) signifies number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a Scale
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
Number analyzed (Participants) | 455 | 1110
score on a Scale | -12.8 (9.73) | 0.2 (9.93)

14. Secondary Outcome: Change From Baseline in Participant-Reported Depressive Symptoms Using the Patient Health Questionnaire - 9 (PHQ-9) Total Score
Description: Change from baseline in PHQ-9 total score were reported. The PHQ-9 was a 9-item, patient-reported outcome measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the Diagnostic and Statistical Manual of Mental Disorders. Each item was rated on a 4-point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses were summed to provide a total score (range of 0 to 27) with higher scores indicating greater severity of depressive symptoms.
Time Frame: IND Phase: Baseline up to 4 weeks; OP/MA Phase: Baseline up to 78 months
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
Number analyzed (Participants) | 453 | 1109
score on a scale | -5.8 (5.84) | 0.6 (6.22)

15. Secondary Outcome: Change From Baseline in Clinical Global Impression-severity (CGI-S) Score
Description: Change from baseline in clinical global impression-severity (CGI-S) score were reported. The CGI-S provides an overall clinician-determined summary measure of the severity of the participant's illness that takes into account all available information, including knowledge of the participant's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participant's ability to function. The CGI-S evaluates the severity of psychopathology on a scale of 1 to 7. Considering total clinical experience, a participant is assessed on severity of mental illness at the time of rating according to: 1 = normal (not at all ill); 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill participants. Negative change in score indicates improvement.
Time Frame: IND Phase: Baseline up to 4 weeks; OP/MA Phase: Baseline up to 78 months
Population: as for outcome 13
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
Number analyzed (Participants) | 456 | 1110
score on a scale | -1.0 [-5.0 to 1] | 0.0 [-5 to 4]

16. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score
Description: Change from baseline in SDS total score were reported. The SDS, a patient-reported outcome measure, was a 5 item questionnaire which had been widely used and accepted for assessment of functional and associated disability impairment. The first three items assessed disruption of (1) work/school, (2) social life, and (3) family life/home responsibilities using a 0-10 rating scale. The score for the first three items were summed to create a total score of 0-30 where a higher score indicated greater impairment.
Time Frame: IND Phase: Baseline up to 4 weeks; OP/MA Phase: Baseline up to 78 months
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
Number analyzed (Participants) | 384 | 1067
score on a scale | -6.4 (7.13) | -0.1 (8.35)

17. Secondary Outcome: Change From Baseline in Participant-Reported Health-related Quality of Life as Assessed by EuroQol-5 Dimension-5 Level (EQ-5D-5L) Valuation Index Score (VAS)
Description: Change from baseline in participant-reported health-related quality of life as assessed by EQ-5D-5L VAS was reported. The EQ-5D-5L is a standardized 2-part instrument for use as a measure of health outcome, primarily designed for self-completion by respondents. It essentially consists of the EQ-5D-5L descriptive system and the EQ-VAS. EQ-VAS self-rating records the respondent's own assessment of his/her overall health status at time of completion, on a scale of 0 (worst health you can imagine) to 100 (best health you can imagine). Positive change in score indicates improvement.
Time Frame: IND Phase: Baseline up to 4 weeks; OP/MA Phase: Baseline up to 78 months
Population: Full analysis set included who received at least 1 dose of intranasal study medication in this study. Here, 'N' (number analyzed) signifies number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
Number analyzed (Participants) | 454 | 1110
score on a scale | 13.0 (18.05) | 0.7 (18.95)

18. Secondary Outcome: Change From Baseline as Assessed by EQ 5D-5L: Sum Score
Description: EQ-5D-5L consists of EQ-5D-5L descriptive system and EQ visual analogue scale (EQ-VAS). EQ-5D-5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "today". Sum score ranges from 0 to 100 where, sum score = (sum of the scores from the 5 dimensions minus 5) *5. Higher score indicates worst health state.
Time Frame: IND Phase: Baseline up to 4 weeks; OP/MA Phase: Baseline up to 78 months
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
Number analyzed (Participants) | 454 | 1110
score on a scale | -10.4 (12.81) | 2.9 (15.88)

19. Secondary Outcome: Change From Baseline in Participant- Reported Health Related Quality of Life Using the Quality of Life in Depression Scale (QLDS)
Description: Change from baseline in participant- reported health related quality of life using the QLDS. The QLDS is a disease-specific validated patient-reported outcome (PRO) measure which assesses the impact that depression has on a participant's quality of life. It is a 34-item self-rated questionnaire which consists of dichotomous response questions, with the response being either True/Not True. Each statement on the QLDS is given a score of "1" or "0". A score of "1" is indicative of adverse quality of life. All item scores are summed to give a total score that ranges from 0 (good quality of life) to 34 (very poor quality of life). A higher score indicates a more severe condition.
Time Frame: IND Phase: Baseline up to 4 weeks; OP/MA Phase: Baseline up to 78 months
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
Number analyzed (Participants) | 293 | 537
score on a scale | -8.2 (8.47) | 0.1 (9.47)

ADVERSE EVENTS:
Time Frame: IND Phase: Baseline up to 4 weeks; OP/MA Phase: Baseline up to 78 months
Description: All enrolled analysis set included all participants who were eligible to enter this study and received at least 1 dose of intranasal study medication.
Arm/Group | Esketamine Nasal Spray (IND Phase) | Esketamine Nasal Spray (OP/MA Phase)
All-Cause Mortality (participants affected / at risk) | 1/458 | 8/1110
Serious Adverse Events (participants affected / at risk) | 5/458 | 212/1110
Other Adverse Events (participants affected / at risk) | 318/458 | 1010/1110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esketamine Nasal Spray (IND Phase) (N=458) | Esketamine Nasal Spray (OP/MA Phase) (N=1110)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 2
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 5
Bradycardia (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 2
Coronary Artery Stenosis (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 4
Pericardial Effusion (Cardiac disorders) | 0 | 1
Myocardial Bridging (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2
Vertigo Positional (Ear and labyrinth disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Duodenal Perforation (Gastrointestinal disorders) | 0 | 1
Gastric Polyps (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Hiatus Hernia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 2
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 2
Pancreatitis Relapsing (Gastrointestinal disorders) | 0 | 1
Umbilical Hernia (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Bile Duct Stone (Hepatobiliary disorders) | 0 | 1
Biliary Obstruction (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 10
Anaphylactic Reaction (Immune system disorders) | 0 | 1
Abscess Limb (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 3
Cellulitis Staphylococcal (Infections and infestations) | 0 | 1
Covid-19 (Infections and infestations) | 0 | 9
Covid-19 Pneumonia (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 0 | 2
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis Salmonella (Infections and infestations) | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 2
Large Intestine Infection (Infections and infestations) | 0 | 1
Necrotising Fasciitis (Infections and infestations) | 0 | 1
Otitis Media Chronic (Infections and infestations) | 0 | 1
Pharyngitis Streptococcal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 7
Postoperative Wound Infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 0 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 3
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 | 1
Animal Bite (Injury, poisoning and procedural complications) | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 2
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Exposure During Pregnancy (Injury, poisoning and procedural complications) | 0 | 1
Face Injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 1
Incisional Hernia (Injury, poisoning and procedural complications) | 0 | 1
Intentional Overdose (Injury, poisoning and procedural complications) | 0 | 3
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 3
Meniscus Injury (Injury, poisoning and procedural complications) | 0 | 2
Multiple Injuries (Injury, poisoning and procedural complications) | 0 | 1
Muscle Rupture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 2
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 2
Blood Pressure Diastolic Increased (Investigations) | 0 | 1
Myocardial Necrosis Marker Increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Obesity (Metabolism and nutrition disorders) | 0 | 1
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Facet Joint Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Anal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Clear Cell Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian Germ Cell Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic Neuroendocrine Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Small Intestine Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Akathisia (Nervous system disorders) | 0 | 1
Carotid Artery Aneurysm (Nervous system disorders) | 0 | 2
Cerebrovascular Accident (Nervous system disorders) | 0 | 2
Dysarthria (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Facial Paralysis (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 3
Hemiparesis (Nervous system disorders) | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 1
Intracranial Aneurysm (Nervous system disorders) | 0 | 2
Ischaemic Stroke (Nervous system disorders) | 0 | 1
Loss of Consciousness (Nervous system disorders) | 0 | 1
Metabolic Encephalopathy (Nervous system disorders) | 0 | 1
Occipital Neuralgia (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Device Breakage (Product Issues) | 0 | 1
Adjustment Disorder (Psychiatric disorders) | 0 | 2
Affect Lability (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 5
Completed Suicide (Psychiatric disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 2
Conversion Disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 18
Depression Suicidal (Psychiatric disorders) | 0 | 1
Major Depression (Psychiatric disorders) | 0 | 3
Mania (Psychiatric disorders) | 0 | 1
Persistent Depressive Disorder (Psychiatric disorders) | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 11
Suicide Attempt (Psychiatric disorders) | 0 | 15
Acute Kidney Injury (Renal and urinary disorders) | 0 | 2
Bladder Outlet Obstruction (Renal and urinary disorders) | 0 | 1
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 6
Renal Artery Stenosis (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Stress Urinary Incontinence (Renal and urinary disorders) | 0 | 2
Urethral Stenosis (Renal and urinary disorders) | 0 | 2
Urge Incontinence (Renal and urinary disorders) | 0 | 1
Urinary Bladder Polyp (Renal and urinary disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 1
Breast Hyperplasia (Reproductive system and breast disorders) | 0 | 1
Cervical Dysplasia (Reproductive system and breast disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 1
Epididymal Cyst (Reproductive system and breast disorders) | 0 | 1
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 0 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 1
Vaginal Prolapse (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vocal Cord Thickening (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abdominoplasty (Surgical and medical procedures) | 0 | 1
Female Sterilisation (Surgical and medical procedures) | 0 | 1
Mammoplasty (Surgical and medical procedures) | 0 | 1
Spinal Fusion Surgery (Surgical and medical procedures) | 0 | 1
Aortic Dissection (Vascular disorders) | 0 | 1
Circulatory Collapse (Vascular disorders) | 0 | 1
Hypertensive Emergency (Vascular disorders) | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Esketamine Nasal Spray (IND Phase) (N=458) | Esketamine Nasal Spray (OP/MA Phase) (N=1110)
Vertigo (Ear and labyrinth disorders) | 77 | 198
Diplopia (Eye disorders) | 15 | 58
Vision Blurred (Eye disorders) | 35 | 116
Abdominal Pain (Gastrointestinal disorders) | 4 | 70
Abdominal Pain Upper (Gastrointestinal disorders) | 6 | 80
Constipation (Gastrointestinal disorders) | 6 | 59
Diarrhoea (Gastrointestinal disorders) | 12 | 184
Hypoaesthesia Oral (Gastrointestinal disorders) | 38 | 83
Nausea (Gastrointestinal disorders) | 82 | 356
Paraesthesia Oral (Gastrointestinal disorders) | 26 | 69
Toothache (Gastrointestinal disorders) | 2 | 84
Vomiting (Gastrointestinal disorders) | 17 | 176
Fatigue (General disorders) | 20 | 145
Feeling Drunk (General disorders) | 25 | 47
Pyrexia (General disorders) | 2 | 84
Bronchitis (Infections and infestations) | 0 | 71
Covid-19 (Infections and infestations) | 0 | 134
Gastroenteritis (Infections and infestations) | 2 | 72
Influenza (Infections and infestations) | 3 | 133
Nasopharyngitis (Infections and infestations) | 13 | 267
Sinusitis (Infections and infestations) | 1 | 74
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 142
Urinary Tract Infection (Infections and infestations) | 7 | 176
Fall (Injury, poisoning and procedural complications) | 1 | 71
Blood Pressure Increased (Investigations) | 35 | 157
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 182
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 226
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 84
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 79
Dizziness (Nervous system disorders) | 95 | 365
Dizziness Postural (Nervous system disorders) | 22 | 57
Dysgeusia (Nervous system disorders) | 77 | 217
Headache (Nervous system disorders) | 70 | 401
Hypoaesthesia (Nervous system disorders) | 44 | 102
Migraine (Nervous system disorders) | 3 | 56
Paraesthesia (Nervous system disorders) | 24 | 92
Sedation (Nervous system disorders) | 25 | 84
Somnolence (Nervous system disorders) | 43 | 253
Anxiety (Psychiatric disorders) | 30 | 197
Depression (Psychiatric disorders) | 1 | 73
Dissociation (Psychiatric disorders) | 100 | 272
Insomnia (Psychiatric disorders) | 16 | 149
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 114
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 23 | 93
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 11 | 95
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 65
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 26 | 60
Hypertension (Vascular disorders) | 1 | 79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT02782104/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT02782104/SAP_001.pdf